CLINICAL TRIAL: NCT00062231
Title: Oral Empirical Therapy of Fever in Low-Risk Neutropenic Cancer Patients: A Prospective, Double-Blind, Randomized, Multicenter Trial Comparing Monotherapy (Single Daily Dose Moxifloxacin) With Combination Therapy (Ciprofloxacin Plus Amoxicillin/Clavulanic Acid)
Brief Title: Moxifloxacin Compared With Ciprofloxacin/Amoxicillin in Treating Fever and Neutropenia in Patients With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: EORTC-46001; EORTC-46001
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Myeloproliferative Disorders; Fever, Sweats, and Hot Flashes; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neutropenia; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: infection; neutropenia; fever, sweats, and hot flashes; unspecified adult solid tumor, protocol specific; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; stage 0 chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; intraocular lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; chronic neutrophilic leukemia; recurrent adult acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Myeloproliferative Disorders; Fever; Hot Flashes; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neutropenia; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin; Moxifloxacin

INTERVENTIONS:
Drug: amoxicillin-clavulanate potassium
Drug: ciprofloxacin
Drug: moxifloxacin hydrochloride
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Antibiotics such as amoxicillin, ciprofloxacin, and moxifloxacin may be effective in preventing or controlling fever and neutropenia in patients with cancer. It is not yet known whether moxifloxacin alone is more effective than amoxicillin combined with ciprofloxacin in treating neutropenia and fever.

PURPOSE: This randomized clinical trial is studying how well moxifloxacin works and compares it to ciprofloxacin together with amoxicillin in treating neutropenia and fever in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rates of successful response to moxifloxacin vs ciprofloxacin in combination with amoxicillin-clavulanate potassium in low-risk febrile neutropenic patients with cancer.
* Compare the time to discharge, time to discontinuation of any antimicrobial therapy, and time to defervescence of patients treated with these regimens.
* Compare 28-day survival of patients treated with these regimens.
* Determine the proportion of these patients who are eligible for oral therapy and a therapeutic management including intention of early discharge.
* Determine the medical and nonmedical reasons for continued in-hospital observation and care or for readmission of these patients.
* Determine the accuracy of the physician's estimate of further neutropenia duration and evaluate its predictive value in these patients.
* Validate the Multinational Association for Supportive Care in Cancer low-risk prediction rule to predict the absence of serious medical complications in the setting of oral therapy in in- and outpatients.

OUTLINE: This is a double-blind, randomized, multicenter study. Patients are stratified according to institution, underlying disease (hematologic malignancy vs other), pretreatment with no more than a single dose (yes vs no), and outpatient status at fever onset (yes vs no). Patients are randomized into 1 of 2 treatment arms.

* Arm I: Patients receive oral moxifloxacin once daily. Patients also receive oral ciprofloxacin placebo and oral amoxicillin-clavulanate potassium placebo twice daily.
* Arm II: Patients receive oral ciprofloxacin and oral amoxicillin-clavulanate potassium twice daily. Patients also receive oral moxifloxacin placebo once daily.

Patients with fever classified as not related to infection (i.e., doubtful) stop antibiotic therapy on day 3. All other patients receive antibiotics until complete resolution of infection, or until failure is determined or anticipated, for up to 28 days.

Patients are followed at 7-10 days.

PROJECTED ACCRUAL: A total of 530 patients (265 patients per treatment arm) will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer with developing febrile neutropenia

  * Neutropenia defined as an absolute granulocyte count of less than 1,000/mm^3, expected to fall to less than 500/mm^3 within 24 hours, secondary to administration of chemotherapy and/or radiotherapy within the past 30 days
  * Fever defined as an oral temperature greater than 38.5ºC once, or 38°C or greater on 2 or more occasions at least 1 hour apart during a 12-hour period, and suspected to be due to infection
* Expected low risk of serious medical complications as predicted by a Multinational Association for Supportive Care in Cancer risk-index score of greater than 20
* No obvious signs of exit-site or tunnel intravascular catheter infection
* No known or suspected CNS infection
* No known or highly suspected bacterial, viral, or fungal infection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* No high probability of death within 48 hours before study enrollment (i.e., patients who are moribund or comatose for any reason with little hope of recovery OR patients in danger of, or in hepatic stupor or coma)

Hematopoietic

* See Disease Characteristics
* No signs or symptoms of uncontrolled bleeding

Hepatic

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* AST and ALT no greater than 5 times ULN
* No severe hepatic dysfunction

Renal

* Creatinine no greater than 3.4 mg/dL
* Creatinine clearance at least 25 mL/min
* No renal failure requiring hemodialysis or peritoneal dialysis

Cardiovascular

* No prior symptomatic arrhythmias
* No clinically relevant bradycardia
* No QTc interval prolongation
* No uncorrected hypokalemia
* No signs or symptoms of hypotension (systolic less than 90 mm Hg)

Pulmonary

* No signs or symptoms of respiratory insufficiency

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to swallow oral medication
* No contraindication for oral drug intake
* No condition likely to severely impair drug absorption
* No prior immediate or accelerated reaction to penicillin, cephalosporin, or fluoroquinolone antibiotics
* No known allergy or hypersensitivity to any antibiotics in this study or other quinolones
* No signs or symptoms of severe dehydration
* No signs or symptoms of shock
* No other signs or symptoms at presentation that would necessitate IV supportive therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* More than 4 days since prior antibacterial agents except for the following:

  * A single (oral or parenteral therapeutic) dose after initial diagnosic work-up and within the last 8 hours
  * Low-dose cotrimoxazole (i.e., no more than 480 mg daily or 960 mg 3 times per week) prophylaxis of Pneumocystis carinii pneumonia
* More than 30 days since prior investigational drugs
* No prior randomization in this study
* No other concurrent antimicrobial agents
* No class IA or class III antiarrhythmic drugs or other concurrent drugs that prolong the QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2002-04; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Response as measured by International Antimicrobial Therapy Group (IATG) specific criteria at the completion of allocated treatment

SECONDARY OUTCOMES:
Rate of complication as measured by Multinational Association for Supportive Care in Cancer (MASCC) criteria at the end of febrile neutropenic episode
Time to discharge as measured by Logrank continuously until the end of febrile neutropenic episode
Time to defervescence as measured by Logrank continuously until the end of febrile neutropenic episode
Survival status as measured by Logrank at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Kern, MD, Study Chair — University Hospital Freiburg
Locations (23):
- Belgium (3):
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
- France (2):
  - Institut Bergonie, Bordeaux
  - Institut Curie Hopital, Paris
- Germany (8):
  - Charite - Campus Charite Mitte, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Klinikum der Albert - Ludwigs - Universitaet Freiburg, Freiburg im Breisgau
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Klinikum der Stadt Mannheim, Mannheim
  - Frauenklinik - Universitaetsklinikum Rostock am Klinikum Sudstadt, Rostock
  - Universitaetsklinikum Ulm, Ulm
- Wolfson Medical Center, Holon, Israel
- Italy (2):
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Universita Degli Studi di Udine, Udine
- Slovakia (2):
  - National Cancer Institute - Bratislava, Bratislava
  - St. Elizabeth Cancer Institute Hospital, Bratislava
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Hopital D'Yverdon, Yverdon-les-Bains
- Turkey (Türkiye) (3):
  - Hacettepe University - Faculty of Medicine, Ankara
  - Ibn-i Sina Hospital, Ankara
  - Marmara University Hospital, Istanbul

REFERENCES:
- [Derived] Kern WV, Marchetti O, Drgona L, Akan H, Aoun M, Akova M, de Bock R, Paesmans M, Viscoli C, Calandra T. Oral antibiotics for fever in low-risk neutropenic patients with cancer: a double-blind, randomized, multicenter trial comparing single daily moxifloxacin with twice daily ciprofloxacin plus amoxicillin/clavulanic acid combination therapy--EORTC infectious diseases group trial XV. J Clin Oncol. 2013 Mar 20;31(9):1149-56. doi: 10.1200/JCO.2012.45.8109. Epub 2013 Jan 28. PMID 23358983